CLINICAL TRIAL: NCT01406951
Title: Diagnostic Value of sTREM-1 and PCT Level as Well as CPIS Score for Ventilator-Associated Pneumonia Among ICU Sepsis Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lixin Xie, Department Of Respiratory Diseases, Chinese PLA General Hospital
Other Study IDs: 301PLAGH-20090923001
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2009-09

CONDITIONS: Sepsis; Ventilator-Associated Pneumonia
Keywords: sTREM-1; PCT; CPIS; VAP; EVC; diagnosis; prognosis
MeSH Terms: conditions — Sepsis; Pneumonia, Ventilator-Associated; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SIRS: (1) temperature > 38oC or < 36oC; (2) pulse rate > 90 beats/min; (3) ventilation rate > 20 breaths/min or hyperventilation with a partial pressure of arterial carbon dioxide (PaCO2) < 32 mmHg; (4) white blood cell (WBC) count >1 2,000μL-1 or < 4000 μL-1 , or > 10% immature cells.
- sepsis: SIRS + infection
- VAP: (1) after 48-72h endotracheal intubation, X-ray film displays new or progressive infiltrating focus; (2)The patient is in two of the following conditions: a. fever (temperature >38 ℃ or higher than basal temperature; b. peripheral WBC count≥10×10∧9/L，or <4×10∧9/L; c. appearance or increase of purulent respiratory tract secretion. Besides the diagnostic norms above, it is suggested that lower respiratory tract secretions be collected under the bronchoscope and half-quantitative etiological culture be carried out through the medium of BALF samples (diagnostic threshold value:104cfu/mL ).

SUMMARY:
Aims: to explore the value of TREM-1 (triggering receptor expressed on myeloid cells-1) ,PCT(Procalcitonin), as well as CPIS (clinical pulmonary infection score) in the diagnostic and prognostic assessment of VAP (ventilator associated pneumonia); and to make a comparison with WBC (white blood cells) and CRP (C-reactive protein) level as well as SOFA (Sequential Organ Failure Assessment) Score Methods: There were 92 subjects of sepsis, who were either receiving endotracheal intubation or had undergone tracheotomy and were exposed to mechanical ventilation. The subjects were divided into the VAP group (32) and the Non-VAP group (60), the criterion being the contraction of VAP 48 hours after ICU admission. Etiological culture was conducted in BALF (bronchoalveolar lavage fluid). And sTREM-1 density was determined by examining serum sTREM-1, PCT, WBC, CRP and EVC (exhaled ventilator condensate). Meanwhile, the CPIS and SOFA score were worked out. With a 28-day survival as the demarcation line, the VAP group was further divided into the survivors group, who stayed alive for 28 days or more , and the non-survivors group, who died within 28 days. The sTREM-1 and PCT level were denoted as meridians (range interquartile), while the WBC and CRP level as well as the CPIS and SOFA score, means±standard deviations (SD).

Results: Averagely, the patients would contract clinically-confirmed VAP 6.9 days after admission, which was mainly traced to Gram-negative bacilli infection. On the very day of diagnosis, compared with the Non-VAP group, the VAP group showed a higher level of serum sTREM-1, PCT, WBC and CRP as well as CPIS and SOFA score（295.6pg/ml vs.143.5pg/ml, P<0.001；4.5ng/ml vs. 1.4ng/ml，P=0.008；16.7×10∧9/L vs.10.9×10∧9/L, P<0.001；11.5mg/dl vs. 7.7mg/dl，P=0.012； 6.0vs. 1.9, P<0.001；10.0vs. 7.5, P=0.017）, AUC (area under the receiver operating characteristic curve）turned out as follows :sTREM-1: 0.73（95% CI 0.61-0.85）;PCT : 0.70（95% CI 0.57-0.83）;WBC: 0.73（95% CI 0.60-0.85）.The CPIS score, which was proved by logistic regression analysis as the sole risky factor to VAP, amounted to 0.96（95% CI 0.91-1.00）. Combined prediction probability containing all the data was calculated in accordance on the relative regression equation. sTREM-1+WBC+CPIS score proved to be most reliable for diagnosis. AUC turned out as 0.98. With 0.277 as the cut-off point, sensitivity measured 0.97, specificity, 0.9 and YDI, 0.87. There were only 5 VAP subjects whose sTREM-1 density could be detected in EVC. The VAP patients were divided into a survivors group (n=15) and a non-survivors group (n=17) with a 28-day survival as the demarcation line. The non-survivors group demonstrated a higher PCT level and higher CPIS & SOFA score than the survivors. （3.0ng/ml vs. 15.3ng/ml，P=0.032；5.4vs. 6.6, P=0.03；8.1vs.11.7 P=0.049). AUC worked out PCT 0.752（95% CI 0.547-0.956）and CPIS 0.764（95% CI 0.575-0.953）. Calculations on the regression equation showed the PCT+CPIS score was most reliable for prognostic assessment. AUC turned out as 0.848. With 0.516 as the demarcation line, sensitivity measured 0.867, specificity, 0.818 and YDI, 0.685.

conclusion: WBC + CPIS helps improve VAP diagnosis; PCT+CPIS may be used for VAP prognostic assessment. Taking two items into consideration will be of guiding value in VAP treatment as well as mortality rate reduction. The sTREM-1 level in EVC，however，may be devoid of value for VAP diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* （1）Male and female aged 18 years old and over;
* （2）Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.（3）Clinically suspected infection; （4）Fulfilled criteria of VAP diagnosis(a) after 48-72h endotracheal intubation, X-ray film displays new or progressive infiltrating focus; (b)The patient is in two of the following conditions: a. fever (temperature >38 ℃ or higher than basal temperature; b. peripheral WBC count≥10×10∧9/L，or <4×10∧9/L; c. appearance or increase of purulent respiratory tract secretion. Besides the diagnostic norms above, it is suggested that lower respiratory tract secretions be collected under the bronchoscope and half-quantitative etiological culture be carried out through the medium of BALF samples (diagnostic threshold value:104cfu/mL ).

Exclusion Criteria:

* (1) were under 18 years of age;
* (2) had contracted VAP upon ICU admission or in less than 48h after being admitted;
* (3) were suffering from acquired immunodeficiency syndrome;
* (4)were suffering from polymorphonuclear granulocyte counts (< 500 μL-1); - (5) died within 24h after being taken into the ICU, or refused to get involved in the study, or gave up treatment during the period of observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between March 2010 and March 2011 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death

CONTACTS AND LOCATIONS:
Overall Officials: Xie Lixin, doctor, Study Director — Department Of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China